CLINICAL TRIAL: NCT02471313
Title: A Pilot Study of an Integrated Imaging Strategy to Phenotype Progression of Liver Tumors During and After Chemoembolization
Brief Title: Integrated Imaging Strategy to Phenotype Progression of Liver Tumors During and After Chemoembolization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 150137; NCT02471313 (Registry Identifier: ClinicalTrials.gov); 15-CC-0137 (Other: NIHCC)
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-03-07

CONDITIONS: Liver Cancer; Liver Neoplasm; Hepatocellular Carcinoma; HCC
Keywords: Cross-Sectional Imaging; Chemoembolization; Radiation Therapy; Tumor Hypoxia; PET Imaging
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- [18F] FMISO PET scan (Experimental): Patients with primary hepatic malignancy who underwent [18F] FMISO PET Scan following transarterial chemoembolization (TACE) procedure
  Interventions: Drug: [18F] FMISO

INTERVENTIONS:
Drug: [18F] FMISO — [18F] Fluromisonidazole, 1 h-(3-[18F]-fluro-2hydroxyl-propy10-2-nitro-imidazaole is an investigational positron emission tomography (PET) radiopharmaceutical for injection and used to visualize hypoxia imaging agent. Each patient will receive up to 10 mCi of [18F] FMISO PET imaging post TACE procedure.
  Other Names: FMISO

SUMMARY:
Background:

- Treatment for liver cancer can include surgery, transplant, and chemotherapy. It can also include other minimally invasive tumor treatments such as transarterial chemoembolization (TACE). TACE treatment for liver cancer helps control the cancer but is not considered a cure. Researchers want to learn more about the effects of TACE on liver tumors and surrounding tissue. To do this, they will use a positive emission test (PET) and a radioactive tracer called [18F] FMISO.

Objectives:

- To see if [18F] FMISO is useful for evaluating what happens to liver tumors and surrounding tissue after TACE.

Eligibility:

- People age 18 and older with liver cancer who have been approved to have TACE.

Design:

* Participants will meet with a study researcher to see if they can take part in the study.
* Participants will have TACE under a separate NCI protocol or at a hospital other than the NIH Clinical Center.
* Before and after TACE, participants will have a CT and MRI of the abdomen. For these scans, they will lie in a machine that takes pictures of their body. They will also have blood tests and a physical exam.
* The [18F] FMISO imaging study will be performed at NIH only.
* Participants will have an intravenous catheter placed in their arm (if they do not have one). The [18F] FMISO tracer will be injected.
* Participants will have PET-CT scans. Each scan will take about 30 minutes.
* Some participants will also have [18F] FMISO and PET-CT scans before TACE.
* As part of standard care for TACE, participants will have CT and MRI scans at regular intervals. This will evaluate tumor response.

DETAILED DESCRIPTION:
Background

* TACE is the standard therapy for inoperable primary liver cancers or tumor control prior to transplantation. The mechanisms for TACE s failure remains poorly understood.
* Although acute hypoxia and significant tumor necrosis occurs following TACE, the tumor adaptive response and localization for such have not been well characterized.
* Imaging tools using a hypoxia-specific tracer [(18)F] FMISO may help identify the pattern and distribution of acute post-TACE tumor hypoxia relative to demonstrated tumor progression.
* The primary hypothesis of this study states that tumor progression post-TACE arises from changes in tumor phenotype induced by treatment-related hypoxia superimposed on the dynamic process of underlying tumor hypoxia.

Objectives

-To determine the feasibility of hypoxic tumor identification despite relatively high liver background signal, and describe patterns of tumor hypoxia in the immediate post-TACE treatment period using PET imaging [(18)F] MISO uptake registered with cross-sectional imaging.

Eligibility

* Patients greater than or equal to 18 years with inoperable primary hepatic malignancy or hepatic-dominant metastatic-disease and be otherwise eligible to receive TACE treatment. Patients with hepatocellular carcinoma should have intermediate stage disease according to the BCLC staging system (Stage A4 or B).
* Patients must not have had chemotherapy- or radiation therapy to liver for at least 2 weeks prior to starting study treatments.
* Patients must not have an acute, critical illness.
* Patients must not be pregnant
* Able to understand and be willing to sign a written informed consent

Design

* Fifteen patients with primary or metastatic liver malignancy will be enrolled into this pilot, non-randomized, open study of the feasibility of using (18)F-fluoromisonidazole PET scanning to determine hypoxic tumor identification and localization, and to identify the pattern and distribution of acute post-TACE tumor hypoxia relative to demonstrated tumor progression.
* Twenty-four to seventy-two hours after standard of care TACE, patients will undergo

PET scanning using 0.1mCi/kg (maximum 10mCi) of (18)F-fluoromisonidazole [(18)F] MISO).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have confirmed inoperable primary hepatic malignancy or hepatic dominant metastatic - neoplastic disease evidenced by histology or cytology, or characteristic enhancement pattern on CT or MRI together with an abnormal serum alpha-fetoprotein >200mg/dl in the case of hepatocellular carcinoma.
* Patients with hepatocellular carcinoma should conform to intermediate stage disease according to the BCLC(16) staging system (Stage A4 or B) and be otherwise eligible to receive TACE treatment.
* Patients must have had no chemotherapy or radiotherapy to the liver therapy for, their malignancy for at least 2 weeks (or until response can be adequately assessed) prior to treatment and must have recovered from all clinically significant side effects of therapeutic and diagnostic interventions.
* Serum creatinine less than or equal to 2.0 mg/dl unless the measured creatinine clearance is greater than 60ml/min
* Age greater than or equal to18 years
* Ability of subject to understand and willingness to sign a written informed consent document
* Patient must be able to lie still for the procedure
* ECOG status less than or equal to 2
* In addition, for patients receiving TACE outside NIH:

  * Patient must have physician willing to collaborate with NIH PI by providing required medical record and digital MR/ CT scan documentation pre and post TACE procedure.
  * Patient must be willing to sign an Authorization for the Release of Medical Information form

EXCLUSION CRITERIA:

* Patients who have received prior TACE treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to misonidazole or other agents used in study.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients of childbearing age must not be pregnant. The effects of [(18)F]FMISO on the developing human fetus are unknown. Pregnancy is a contraindication for TACE.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06-12; Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot B Levy, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] THOMLINSON RH, GRAY LH. The histological structure of some human lung cancers and the possible implications for radiotherapy. Br J Cancer. 1955 Dec;9(4):539-49. doi: 10.1038/bjc.1955.55. No abstract available. PMID 13304213
- [Background] Vaupel P, Mayer A, Hockel M. Tumor hypoxia and malignant progression. Methods Enzymol. 2004;381:335-54. doi: 10.1016/S0076-6879(04)81023-1. No abstract available. PMID 15063685
- [Background] Durand RE, Aquino-Parsons C. Non-constant tumour blood flow--implications for therapy. Acta Oncol. 2001;40(7):862-9. doi: 10.1080/02841860152703508. PMID 11859987
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-CC-0137.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | [18F] FMISO PET Scan
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [18F] FMISO PET Scan
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Transarterial Chemoembolization procedure [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which Uptake of [18F]-FMISO Was Successful and Hypoxic Tumors Were Observed During PET Scan Imaging Post TACE Procedure
Description: A single dose of study imaging agent [18F] FMISO was administered following the TACE procedure. PET Scan imaging was then performed to evaluate if hypoxic tumor identification were observable following administration of study imaging agent. Power and significance calculations are not applicable to this small sample feasibility study.
Time Frame: up to 72 hours after injection of [18F] FMISO
Measure: Count of Participants; unit: Participants
Groups:
- Uptake of [18F] FMISO With PET Scan Imaging: Patients with primary hepatic malignancy who underwent [18F] FMISO PET Scan following transarterial chemoembolization (TACE) procedure
  [18F] FMISO: [18F] Fluromisonidazole, 1 h-(3-[18F]-fluro-2hydroxyl-propy10-2-nitro-imidazaole is an investigational positron emission tomography (PET) radiopharmaceutical for injection and used to visualize hypoxia imaging agent. Each patient will receive up to 10 mCi of [18F] FMISO PET imaging post TACE procedure.
Arm/Group | Uptake of [18F] FMISO With PET Scan Imaging
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected within 24 hours post [18F] FMISO injection on all study participants
Groups:
- [18F] FMISO PET Scan: Patients with primary hepatic malignancy are undergo [18F] FMISO PET Scan following transarterial chemoembolization (TACE) procedure.
Arm/Group | [18F] FMISO PET Scan
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [18F] FMISO PET Scan (N=3)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT02471313/Prot_SAP_000.pdf